CLINICAL TRIAL: NCT00689533
Title: VEPTR Implantation to Treat Children With Early Onset Scoliosis Without Rib Abnormalities: a Prospective Multicenter Study
Brief Title: VEPTR Implantation to Treat Children With Early Onset Scoliosis Without Rib Abnormalities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Chest Wall and Spine Deformity Research Foundation (Other)
Responsible Party: Study Group Coordinator, Chest Wall and Spine Deformity Study Group
Other Study IDs: CWSD0003
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Congenital Progressive Scoliosis; Infantile
Keywords: VEPTR; TIS; scoliosis; juvenile
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Objective: To evaluate the use of unilateral or bilateral VEPTR devices, with or without expansion thoracoplasty, for preventing further progression of the Cobb angle, allowing for spinal growth and improving pulmonary function in the treatment of children with progressive scoliosis without rib abnormalities.

DETAILED DESCRIPTION:
Number of Patients Planned: A total of 250 patients requiring treatment with the VEPTR device and meeting the inclusion/exclusion criteria will be enrolled in the study. All patients enrolled in this study will receive the VEPTR device.

Duration of Follow-up: Patients will be clinically followed post-surgery throughout the course of the patient's treatment. Follow-up appointments will be scheduled at 1, 6, and 12 months post-surgery and every year thereafter until 5 years after the index procedure, then every 2 years until the final planned procedure, or the completion or spinal growth (typically about 2 years after menarche in girls, or the equivalent in boys), whichever occurs first. Other patient visits may occur as deemed necessary.

General Design and Methodology: This is a prospective, multi-center, clinical study to evaluate the use of VEPTR devices for preventing further progression of the Cobb angle, a measure of the curvature of the spine, determined from measurements made on radiographs, allowing for spinal growth and improving pulmonary function in the treatment of children with progressive scoliosis without rib abnormalities. Unilateral vs. Bilateral, and use of an opening wedge thoracostomy, are at the discretion of the surgeon. The treatment would be used regardless of the study, therefore it is routine care. The primary study hypothesis is that, in regard to key clinical and radiographic outcomes, the success rate of the VEPTR device is at least 90%. A secondary study hypothesis is that in regards to key pulmonary outcomes (improvement in pulmonary function tests and increase in lung volume as measured by CT scans), the success rate of the VEPTR device is at least 90% (see Primary Study Endpoints below). Details of the patient outcomes and the study hypothesis are given below. With correction for 10% attrition, 250 patients split between the participating institutions will be enrolled.

Primary Study Endpoints: The primary endpoint will be based on the findings up to and including the last scheduled patient follow-up visit. An individual patient's treatment will be considered successful only if each of the following criteria are met:

* The patient's Cobb angle at the final surgery is less than or equal to the patient's pre-operative Cobb angle and
* The patient's trunk height or spinal length at final surgery is greater than or equal to the patient's immediate post-operative trunk height or spinal length

ELIGIBILITY:
Inclusion Criteria:

* Progressive scoliosis: idiopathic, congenital, syndromic, neuromuscular
* Progressive scoliosis with a Cobb angle that has advanced beyond 45˚
* 18 months to 10 years of age with open triradiate cartilages

Exclusion Criteria:

* Presence of fused ribs
* Presence of multiple absent ribs
* Thoracic dysplasia such as Jeune's syndrome or equivalent condition
* Prior spinal fusion or spinal instrumentation
* Patient is participating in another clinical trial using investigational devices/drugs
* Patient is unable or unwilling to sign a consent form

Ages: 18 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be selected from participating children's hospitals, most likely during spine clinic.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The patient's Cobb angle at the final surgery is less than or equal to the patient's pre-operative Cobb angle | Anticipate 6 years
The patient's trunk height or spinal length at final surgery is greater than or equal to the patient's immediate post-operative trunk height or spinal length | Anticipate 6 years

CONTACTS AND LOCATIONS:
Overall Officials: John M Flynn, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Shriners Hospital for Children, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah